CLINICAL TRIAL: NCT04880980
Title: Comparison of Efficacy of Double Dose Oral Terbinafine Versus Itraconazole in Treatment of Dermatophyte Infections of Skin - A Prospective, Randomized Controlled Trial
Brief Title: Comparison of Efficacy of Double Dose Oral Terbinafine Vs Itraconazole in Treatment of Dermatophyte Infections of Skin.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pak Emirates Military Hospital (Other)
Responsible Party: Principal Investigator, Dr. Umar Abdul Ali Qureshi, Speciality Registrar Dermatology, Pak Emirates Military Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PEMH Rawalpindi
Record Dates: First submitted 2021-03-16; First posted 2021-05-11 (Actual); Last update posted 2022-04-01 (Actual); Status verified 2022-03

CONDITIONS: Dermatophyte Infection; Terbinafine Adverse Reaction; Itraconazole Adverse Reaction
Keywords: double dose; oral terbinafine; oral itraconazole; dermatophyte skin infection; randomized controlled trial
MeSH Terms: conditions — Dermatomycoses | interventions — Terbinafine; Itraconazole; icon infiltrant

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Who Masked: Participant
Masking Description: Participants will be randomly assigned to group one or two.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Efficacy of double dose oral terbinafine in treatment of dermatophytic infections of skin (Active Comparator): This group of participants will be given double than usual dose of oral terbinafine for the treatment of dermatophyte skin infections.
  Interventions: Drug: Terbinafine Pill
- Efficacy of double dose oral itraconazole in treatment of dermatophytic infections of skin (Active Comparator): This group of participants will be given double than usual dose of oral itraconazole for the treatment of dermatophyte skin infections
  Interventions: Drug: Itraconazole capsule

INTERVENTIONS:
Drug: Terbinafine Pill — Double than usual dose of oral terbinafine pills will be used for treatment purpose in one group.
  Other Names: Lamisil
  Arms: Efficacy of double dose oral terbinafine in treatment of dermatophytic infections of skin
Drug: Itraconazole capsule — Double than usual dose of oral itraconazole capsules will be used for treatment purpose in second group.
  Other Names: Icon
  Arms: Efficacy of double dose oral itraconazole in treatment of dermatophytic infections of skin

SUMMARY:
Study would be conducted to compare the efficacy and safety of double than usual dose oral terbinafine versus itraconazole in treatment of dermatophyte infections of skin in patient presenting at dermatology department of Pak Emirates Military Hospital, Rawalpindi, Pakistan.

DETAILED DESCRIPTION:
* Study would be a randomized controlled trial, in which 120 subjects would be randomly divided into two equal groups of 60 each.
* Each group would be prescribed double than usual dose of terbinafine(250 mg twice daily) or itraconazole(100mg twice daily) for 2 weeks initially. Treatment may be extended to 4 weeks if cure has not been achieved.

Patients will be diagnosed and followed on the basis of classical clinical features of dermatophyte infections and microscopic potassium hydro-oxide slide preparation for fungal hyphae and spores.

Liver function tests will be checked on day 0, 14 and 28. Individuals aged 15-50 years with one or no co-morbidity will be included in the study.

Study will be conducted over a period of 6-8 months.

ELIGIBILITY:
Inclusion Criteria:

* individuals with dermatophyte skin infection, aged 15-50 years with one or no co-morbidities.

Exclusion Criteria:

* individuals with two or more co-morbidities or known cases of chronic liver disease.

Ages: 15 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 120 (Actual)
Dates: Start 2021-03-15 (Actual); Primary Completion 2022-03-15 (Actual); Study Completion 2022-03-15 (Actual)

PRIMARY OUTCOMES:
Percentage of patients cured by using double dose of oral terbinafine Vs itraconazole in the treatment of resistant dermatophyte skin infections as assessed by measuring pruritis, erythema and scaling . | 2-4 weeks
  Classical clinical features of dermatophyte skin infections (pruritis, erythema and scaling, all will be graded on a scale 0-3 i. e 0=none to 3=severe) would be noted at start of treatment after 2 weeks and then if required after 4 weeks of treatment.
Adverse effects including effects on liver function tests of double dose oral terbinafine Vs itraconazole in the treatment of resistant dermatophyte skin infections. | 2-4 weeks
  Objective Assessment of adverse effects (nausea, vomiting, jaundice) as well as laboratory evaluation of liver function tests (Bilirubin umol/L, ALT U/L, ALP U/L) would be performed at start of treatment after 2 weeks and if required than after 4 weeks.

SECONDARY OUTCOMES:
Duration of treatment required to achieve cure from resistant dermatophyte infections. | 2-4 weeks
  Treatment response in form of clinical features (changes in erythema. Pruritis and scaling) and KOH fungal slide smear testing would be done after 2 weeks of treatment and if required than after 4 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Umar Abdul Ali Qureshi, MBBS, Principal Investigator — Pak Emirates Military Hospital
Locations (1):
- Pak Emirates Military Hospital, Rawalpindi, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No
Individual participant's data will be kept confidential.